CLINICAL TRIAL: NCT04886206
Title: Phase I Study Testing the Injection of Lymphocytes From Haplo-identical Donor Following Chemotherapy in Patients With High-risk Acute Myeloblastic Leukemia Not Eligible for an Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Injection of Lymphocytes From Haplo-identical Donor Following Chemotherapy in Patients With High-risk Acute Myeloblastic Leukemia Not Eligible for an Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: ILDA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC20_0357
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Continual Reassessment Method for MTD
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: DLI — the patients will receive the injection of donor lymphocytes from haplo-identical donor (the son or daughter or possibly nephew or niece of the patient). No immunosuppressive drugs will be used. The HLI dose levels are 1) 1x107 CD3+/kg 2) 5x107 CD3+/kg 3) 7.5x107 CD3+/kg 4) 1x108 CD3+/kg.The CRM method (Continual Reassessment Method) was chosen to specify the dose of cells to be injected, each patient being assigned a dose that is believed to be associated with the target toxicity corresponding to the maximum tolerated dose (MTD). The dose-toxicity curve will be readjusted after assessing the toxicity of each patient.

SUMMARY:
Patients with high risk AML non eligible for an intensive treatment and for an allogeneic transplantation will be treated with azacitidine and venetoclax. The fourth, fifth and sixth injection of azacitidine will be followed by injection of haplo-identical lymphocytes (HLI). This is a single-center phase I study to identify the dose of HLI with the most tolerable toxicity. TheBayesian continuous reassessment method (CRM) will be used

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* patients with de novo or secondary AML, with an unfavorable or intermediate karyotype (according to the 2017 ELN classification), or patients with relapsing AML who may receive second-line treatment
* not candidates for intensive induction, for the following reasons

  * 75 years or ≥ 18 to 74 years and at least one of the following comorbidities: PS ≥ 2 or a history of heart failure requiring treatment or LVEF ≤ 50% or chronic stable angina or FEV1 ≤ 65% or DLCO ≤ 65% or creatinine clearance <45 ml / min; or liver damage with total bilirubin> 1.5 N or other comorbidities that the hematologist considers incompatible with intensive treatment
* ineligible for a classic allogeneic hematopoietic stem cell transplant due to the presence of co-morbidities or too high a risk of toxicity >70 years old or at least one of the following comorbidities: PS ≥ 2 or a history of heart failure requiring treatment or LVEF ≤ 50% or chronic stable angina or FEV1 ≤ 65% or DLCO ≤ 65% or creatinine clearance <45 ml / min; or liver damage with total bilirubin> 1.5 N
* may receive chemotherapy with hypomethylating agents have a partially compatible (haplo-identical) major family donor (≥18 years old) eligible for lymphocyte donation.

Exclusion Criteria:

* AML with favorable karyotype (according to ELN 2017) in RC1
* Patient with refractory or progressive AML
* Other progressive cancer in progress
* Karnosky index <60% or PS> 2
* Severe hepatic function disturbance: transaminases> 5 N, hyperbilirubinemia> 30 µm / L
* Severe infection requiring hospitalization.
* Psychiatric illness compromising the understanding of the information or the carrying out of the study.
* woman of childbearing potential and refusing an effective method of contraception.
* Minor
* Adult under tutorship or curatorship, under legal protection or under family authorization
* Minor family donor (<18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
number of DLT | by day 14

SECONDARY OUTCOMES:
cumulative incidence of relapse | 1 YEAR
relapse-free survival | 1 YEAR
overall survival | 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Guillaume, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France